CLINICAL TRIAL: NCT04998617
Title: Effects of Curcumin-containing Toothpaste on Dental Biofilm and Associated Oral Halitosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 20-3428
Record Dates: First submitted 2021-08-05; First posted 2021-08-10 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Halitosis
MeSH Terms: conditions — Halitosis | interventions — Toothpastes; Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Toothpaste Containing Curcumin (Experimental): After screening, participants will be randomly assigned to receive toothpaste that contains 0.5% curcumin.
  Interventions: Other: Toothpaste with curcumin
- Toothpaste Without Curcumin (Placebo Comparator): After screening, participants will be randomly assigned to receive toothpaste that does not contain curcumin.
  Interventions: Other: Toothpaste without curcumin

INTERVENTIONS:
Other: Toothpaste with curcumin — Subjects will be given toothpaste to be used during this study with 0.5% curcumin
  Arms: Toothpaste Containing Curcumin
Other: Toothpaste without curcumin — Subjects will be given toothpaste to be used during this study without curcumin
  Arms: Toothpaste Without Curcumin

SUMMARY:
Purpose: To investigate the short-term clinical effect of curcumin-containing toothpaste on halitosis as compared to placebo and to assess potential shifts in the composition of dental biofilm associated with the use of curcumin-containing toothpaste

Participants: This clinical study will 30 adult participants under prophylactic or periodontal maintenance protocol.

Procedures (methods): Participants will be included and throughout the protocol will not allow the use any other oral hygiene products except standard manual toothbrush and study toothpaste (either test -curcumin-containing or placebo). Additionally participants will be instructed to odiferous foods such as onions, garlic and spices. At each of the three examination sessions, Plaque Index (six sites, O'Leary) and volatile sulphur compounds (VSC) will be measured.

ELIGIBILITY:
Inclusion Criteria

* Participants must be adult males or females between the ages of 18 and 65 years (inclusive) reporting halitosis
* Participants must be able and willing to follow study procedures and instructions
* Participants must have read, understood and signed an informed consent form
* Participants must present with at least 8 teeth in the functional dentition and with at least 4 teeth in each posterior sextant, 3 of which are adjacent teeth with interproximal papilla in each posterior sextant that will have the stent
* Participants must be in good general health

Exclusion Criteria

* Patients ongoing restorative or periodontal dental treatment or any other medical treatment
* Subjects with any pathological alterations of the oral mucosa
* Any known allergy to previously used oral hygiene products or any known allergy to any of the ingredients of the study products, which are used during the study
* Pregnant women
* Subjects with untreated periodontitis or active caries lesion
* Subjects diagnosed with acute sinusitis, bronchitis or tonsillitis
* Subjects under treatment on medications which can cause malodor, e.g. amphetamines, nitrates and nitrites
* Known diabetes, liver or kidney insufficiency
* Subjects diagnosed with reduced salivary flow due to pathological reasons (e.g. Sjögren syndrome)
* Subjects who underwent preventive periodontal treatment, i.e. oral prophylaxis treatment, within the last week
* Volunteers unwilling to abstain from additional oral hygiene (only tooth brushing allowed) particularly mouthrinse, chewing gums, breath strips, etc and alcohol 12 h prior the first measurement at the study site and until the completion of all measurements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Volatile Sulphur Compounds (VSC) at day 7 | day 7
  Volatile Sulphur Compounds (VSC) values for all subjects will be recorded. F-tests will be used to compare the curcumin group with the placebo group at each timepoint. P-values less than 0.05 will be considered statistically significant. Analyses will be performed using SAS Version 9.4 (SAS Institute, Cary NC).
Volatile Sulphur Compounds (VSC) at day 14 | day 14
  Volatile Sulphur Compounds (VSC) values for all subjects will be recorded. F-tests will be used to compare the curcumin group with the placebo group at each timepoint. P-values less than 0.05 will be considered statistically significant. Analyses will be performed using SAS Version 9.4 (SAS Institute, Cary NC).
Volatile Sulphur Compounds (VSC) at day 21 | day 21
  Volatile Sulphur Compounds (VSC) values for all subjects will be recorded. F-tests will be used to compare the curcumin group with the placebo group at each timepoint. P-values less than 0.05 will be considered statistically significant. Analyses will be performed using SAS Version 9.4 (SAS Institute, Cary NC).
Repeated Measures Regression of Volatile Sulphur Compounds (VSC) | baseline, 21 days
  A repeated measures regression with VSC as the response and treatment (curcumin or negative control) and time (7, 14 or 21 days) as predictors. An autoregressive correlation matrix will be used to account for the correlation between repeated measures within subject.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Moretti, DDS, MS, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: 9 to 36 months following publication
Access Criteria: The investigator who proposes to use the data has approval from an IRB, IEC, or REB and an executed data use/sharing agreement with UNC.